CLINICAL TRIAL: NCT05298657
Title: The Angiotensin-Melatonin Axis in Poor and Hyper Responders for IVF Treatment
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fatima College of Health Sciences (Other)
Collaborators: ART Fertility Clinics LLC (Other)
Responsible Party: Principal Investigator, Rym Ghimouz, Assistant Professor of Biology, Fatima College of Health Sciences
Other Study IDs: FCEC-1-21-22-GRD-1-SF; REFA073 (Other: ART Fertility Clinic Middle East Ethical Approval)
Record Dates: First submitted 2022-03-17; First posted 2022-03-28 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-07

CONDITIONS: Poor Response to Ovulation Induction; PCOS; Endometriosis; Infertility, Female
MeSH Terms: conditions — Endometriosis; Infertility, Female

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Weeks
Biospecimen Retention: Samples Without DNA — Urine samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Poor IVF Treatment Responders
- Hyper IVF Treatment Responders
- Normal responders/ Control group

SUMMARY:
According the World Health Organization (WHO), infertility is a disease of the male or female reproductive system defined by the failure to achieve a pregnancy after 12 months or more of regular unprotected sexual intercourse. In-vitro-fertilization (IVF) is considered to be a successful tool to overcome infertility. However, the current methods used to assess the ovarian reserve and to develop an optimal individualized controlled ovarian hyperstimulation (COH) protocol have shown some limitations. Growing evidence indicates that altered renal renin-angiotensin system (RAS) and/or melatonin are linked to infertility. Aims and Objectives: The current 2 years duration study aims first to investigate the demographic and clinical profiles of patients undergoing IVF in the UAE. In the second phase of the study, we hypothesis that an altered angiotensin-melatonin axis may be considered as an unfavorable prognosis factor in poor and hyper responders undergoing IVF treatment. This hypothesis will be assessed using an observational, longitudinal, prospective clinical study to determine whether the urinary angiotensinogen and/or melatonin deficiency might be present in poor and hyper responders undergoing IVF treatment. Thus, negatively impacting the clinical pregnancy rate. Methodology: various patient's data will be collected using a questionnaire and the levels of angiotensinogen and melatonin in patient's urine will be measured using ELISA test prior to, during and after the IVF treatment. To determine whether the angiotensinogen-melatonin axis disruption affects the IVF treatment outcome, we will analyze the following parameters: the AMH, Antral Follicular Count (AFC), day 2-4 FSH levels, the stimulation cycle in regards to number of stimulation days and amount of gonadotropins used for stimulation, number of oocytes retrieved and number of mature oocytes, quality and embryo's ploidy, number of available euploid embryos and the clinical pregnancy rate after frozen embryo transfer.

DETAILED DESCRIPTION:
Infertility affects approximately 1 in every 4 couples and the WHO (World Health Organization) has defined infertility as a "disease" (World Health Organization (WHO). International Classification of Diseases, 11th Revision (ICD-11) Geneva: WHO 2018.). Rates of infertility are expected to increase in the future as many couples tend to postpone family planning due to various reasons (Mills et al., 2011). Assisted Reproductive Techniques (ART), with In-vitro-fertilization (IVF) being a part of the treatment options, are a successful tool to overcome infertility (Franasiak & Scott, 2014). However, more research to thwart the global burden of infertility is required. This is possible if the underlying causes of infertility can be identified, and personalized therapy implemented (Sun et al., 2019).

Poor and hyper responders are a diverse group of IVF patients, with specific needs. Their management can help in increasing the clinical pregnancy rates. Identifying and understanding how the endocrine variants are linked to the success of IVF responsiveness may lead to a better treatment strategy aimed at achieving successful live births.

Growing evidence indicates that altered renal renin-angiotensin system (RAS) and melatonin are linked to infertility, PCOS and endometriosis.

According to the literature, hyperandrogenemia in an experimental rat model of PCOS has been associated with an upregulation of the intrarenal RAS (Torres Fernandez et al. 2019). When compared to the eutopic endometrium in the proliferative phase, patients with endometriotic cysts had a significant increase in the expression of angiotensin type AT1 and AT2 receptors. This suggests that RAS may be involved in the pathophysiology of endometriosis (Nakao et al. 2017; Nakajima et al. 2018). In addition, alterations in the expression of Angiotensin-converting enzyme, ACE-1, ACE-2, and ACE-3 might be one of the most important mechanisms underlying both female and male infertility (Chen, Bi, Su, Chappell, & Rose, 2016; Pan, Zhan, Le, Zheng, & Jin, 2013).

On the other hand, the levels of melatonin, a powerful antioxidant and an effective free radical scavenger that protects ovarian follicles during follicular maturation are increasing in preovulatory follicular fluid and seem to have an important role in ovulation (Tamura et al., 2012). Similarly, melatonin requirements appear to increase during pregnancy (Voiculescu, Zygouropoulos, Zahiu, & Zagrean, 2014). Melatonin levels are found to be lower in patients with PCOS (Mojaverrostami et al. 2019). And several studies suggest a potential link between melatonin and endometriosis (Mosher et al. 2019; Anderson 2019), leading to the use of melatonin as an adjuvant in the treatment of endometriosis (Mosher et al. 2019; Yesildaglar et al. 2016).

Clinical hypothesis:

This observational, longitudinal, prospective clinical study will investigate the IVF population demographic and clinical profile in the UAE. It will also test the hypothesis whether an altered angiotensin-melatonin axis may be considered an unfavorable prognosis factor in poor responders with or without endometriosis and hyper (PCOS) responders undergoing IVF treatment. Thus, negatively impacting the clinical pregnancy rate.

ELIGIBILITY:
Inclusion Criteria:

depending on the ART Fertility Clinic patients, we are intending to include:

1. Women diagnosed with infertility (when pregnancy is not achieved after 1 year of having regular sexual intercourse without birth control for those under 35 years of age or if pregnancy is not achieved after 6 months of trying to conceive naturally for those older than 35 years of age). Further on, women with proven tubal factor infertility or couples with infertility as a result of a male factor, without the previously mentioned time of not achieving a pregnancy.
2. Women undergoing or in the way to undergo IVF and classified as poor responders according to the four groups of the POSEIDON criteria (Conforti et al., 2019), including patients with a previous oral contraceptive intake.
3. Women diagnosed with PCOS based on the Rotterdam criteria (Rotterdam ESHRE/ASRM-Sponsored PCOS Consensus Workshop Group, 2004.
4. Women diagnosed with endometriosis confirmed by Laparoscopy or visible endometrioma without being diagnosed by laparoscopy (If possible to be enrolled in the research).
5. Women planned to undergo IVF treatment and categorized as expected normal responders) (Ozkan, 2019).
6. Patients under thyroid medication.

Exclusion Criteria:

1. Presence or history of endocrine abnormalities (at the exception of patients who are under thyroid medication).
2. Abnormal outcome of blood biochemistry or hematology.
3. Obese patients with BMI > 40.
4. Couples for whom the male partner has to undergo surgical sperm retrieval.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: From the ART Fertility Clinic, Abu Dhabi, UAE, our collaborator in the project, we are planning to enroll (following the selection criteria detailed below) for a duration of 18 months, IVF female patients aged between 18 and 45 years old and who volunteer to participate in the study. Participants in the study have to sign a participant Information sheet and consent form specific to the urine testing before their enrollment in the study. A questionnaire will be filled out with the different demographics and a summary of the IVF protocol details.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Differences on urine levels of angiotensinogen-melatonin-creatinine ratio between two groups: one with AMH < 1.1 ng/ml against other with AMH > 6.25 ng/ml. | 18 months
  Urinary excretion of angiotensinogen will be analyzed by sandwich-ELISA assay. Urinary melatonin excreted overnight will be determined through the 6-sulfatoxymelatonin molecule. This is a metabolite released in the urine that correlates directly with the melatonin produced, being a noninvasive method of dosing the said molecule. The urinary dosage of 6-sulfatoximelatonin will be performed by the ELISA technique according to the manufacturer's recommendations (IBL International Germany). All molecules will be quantitated using ELISA according to supplier's specifications.

CONTACTS AND LOCATIONS:
Overall Officials: Rym Ghimouz, PhD, Principal Investigator — Fatima College of Health Sciences; Barbara Lawrenz, PhD, Principal Investigator — ART Fertility Clinics; Luciana Campos, PhD, Principal Investigator — Universidade Anhembi Morumbi
Locations (1):
- ART Fertility Clinic, Abu Dhabi, Abu Dhabi Emirate, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anderson G. Endometriosis Pathoetiology and Pathophysiology: Roles of Vitamin A, Estrogen, Immunity, Adipocytes, Gut Microbiome and Melatonergic Pathway on Mitochondria Regulation. Biomol Concepts. 2019 Jul 19;10(1):133-149. doi: 10.1515/bmc-2019-0017. PMID 31339848
- [Background] Barbakadze L, Kristesashvili J, Khonelidze N, Tsagareishvili G. The correlations of anti-mullerian hormone, follicle-stimulating hormone and antral follicle count in different age groups of infertile women. Int J Fertil Steril. 2015 Jan-Mar;8(4):393-8. doi: 10.22074/ijfs.2015.4179. Epub 2015 Feb 7. PMID 25780521
- [Background] Chen K, Bi J, Su Y, Chappell MC, Rose JC. Sex-Specific Changes in Renal Angiotensin-Converting Enzyme and Angiotensin-Converting Enzyme 2 Gene Expression and Enzyme Activity at Birth and Over the First Year of Life. Reprod Sci. 2016 Feb;23(2):200-10. doi: 10.1177/1933719115597760. Epub 2015 Aug 4. PMID 26243544
- [Background] Conforti A, Esteves SC, Cimadomo D, Vaiarelli A, Di Rella F, Ubaldi FM, Zullo F, De Placido G, Alviggi C. Management of Women With an Unexpected Low Ovarian Response to Gonadotropin. Front Endocrinol (Lausanne). 2019 Jun 27;10:387. doi: 10.3389/fendo.2019.00387. eCollection 2019. PMID 31316461
- [Background] Franasiak JM, Scott RT Jr. Embryonic aneuploidy: overcoming molecular genetics challenges improves outcomes and changes practice patterns. Trends Mol Med. 2014 Sep;20(9):499-508. doi: 10.1016/j.molmed.2014.06.006. Epub 2014 Aug 8. PMID 25113799
- [Background] Irani M, Robles A, Gunnala V, Reichman D, Rosenwaks Z. Optimal parameters for determining the LH surge in natural cycle frozen-thawed embryo transfers. J Ovarian Res. 2017 Oct 16;10(1):70. doi: 10.1186/s13048-017-0367-7. PMID 29037231
- [Background] Kuwayama M. Highly efficient vitrification for cryopreservation of human oocytes and embryos: the Cryotop method. Theriogenology. 2007 Jan 1;67(1):73-80. doi: 10.1016/j.theriogenology.2006.09.014. Epub 2006 Oct 20. PMID 17055564
- [Background] La Marca A, Sunkara SK. Individualization of controlled ovarian stimulation in IVF using ovarian reserve markers: from theory to practice. Hum Reprod Update. 2014 Jan-Feb;20(1):124-40. doi: 10.1093/humupd/dmt037. Epub 2013 Sep 29. PMID 24077980
- [Background] Levi-Setti PE, Zerbetto I, Baggiani A, Zannoni E, Sacchi L, Smeraldi A, Morenghi E, De Cesare R, Drovanti A, Santi D. An Observational Retrospective Cohort Trial on 4,828 IVF Cycles Evaluating Different Low Prognosis Patients Following the POSEIDON Criteria. Front Endocrinol (Lausanne). 2019 May 8;10:282. doi: 10.3389/fendo.2019.00282. eCollection 2019. PMID 31139146
- [Background] Mills M, Rindfuss RR, McDonald P, te Velde E; ESHRE Reproduction and Society Task Force. Why do people postpone parenthood? Reasons and social policy incentives. Hum Reprod Update. 2011 Nov-Dec;17(6):848-60. doi: 10.1093/humupd/dmr026. Epub 2011 Jun 7. PMID 21652599
- [Background] Mojaverrostami S, Asghari N, Khamisabadi M, Heidari Khoei H. The role of melatonin in polycystic ovary syndrome: A review. Int J Reprod Biomed. 2019 Dec 30;17(12):865-882. doi: 10.18502/ijrm.v17i12.5789. eCollection 2019 Dec. PMID 31970309
- [Background] Mosher AA, Tsoulis MW, Lim J, Tan C, Agarwal SK, Leyland NA, Foster WG. Melatonin activity and receptor expression in endometrial tissue and endometriosis. Hum Reprod. 2019 Jul 8;34(7):1215-1224. doi: 10.1093/humrep/dez082. PMID 31211323
- [Background] Nakajima T, Chishima F, Nakao T, Hayashi C, Kasuga A, Shinya K, Nakayama T, Azuma H, Ichikawa G, Komatsu A, Yamamoto T, Kawana K. The Expression of MAS1, an Angiotensin (1-7) Receptor, in the Eutopic Proliferative Endometria of Endometriosis Patients. Gynecol Obstet Invest. 2018;83(6):600-607. doi: 10.1159/000490561. Epub 2018 Jul 6. PMID 29982252
- [Background] Nakao T, Chishima F, Sugitani M, Tsujimura R, Hayashi C, Yamamoto T. Expression of Angiotensin II Types 1 and 2 Receptors in Endometriotic Lesions. Gynecol Obstet Invest. 2017;82(3):294-302. doi: 10.1159/000447591. Epub 2016 Jul 7. PMID 27384958
- [Background] Pan PP, Zhan QT, Le F, Zheng YM, Jin F. Angiotensin-converting enzymes play a dominant role in fertility. Int J Mol Sci. 2013 Oct 21;14(10):21071-86. doi: 10.3390/ijms141021071. PMID 24152441
- [Background] Rotterdam ESHRE/ASRM-Sponsored PCOS Consensus Workshop Group. Revised 2003 consensus on diagnostic criteria and long-term health risks related to polycystic ovary syndrome. Fertil Steril. 2004 Jan;81(1):19-25. doi: 10.1016/j.fertnstert.2003.10.004. PMID 14711538
- [Background] Rubio C, Rodrigo L, Garcia-Pascual C, Peinado V, Campos-Galindo I, Garcia-Herrero S, Simon C. Clinical application of embryo aneuploidy testing by next-generation sequencing. Biol Reprod. 2019 Dec 24;101(6):1083-1090. doi: 10.1093/biolre/ioz019. PMID 30721942
- [Background] Steiner AZ, Pritchard D, Stanczyk FZ, Kesner JS, Meadows JW, Herring AH, Baird DD. Association Between Biomarkers of Ovarian Reserve and Infertility Among Older Women of Reproductive Age. JAMA. 2017 Oct 10;318(14):1367-1376. doi: 10.1001/jama.2017.14588. PMID 29049585
- [Background] Sun H, Gong TT, Jiang YT, Zhang S, Zhao YH, Wu QJ. Global, regional, and national prevalence and disability-adjusted life-years for infertility in 195 countries and territories, 1990-2017: results from a global burden of disease study, 2017. Aging (Albany NY). 2019 Dec 2;11(23):10952-10991. doi: 10.18632/aging.102497. Epub 2019 Dec 2. PMID 31790362
- [Background] Tamura H, Takasaki A, Taketani T, Tanabe M, Kizuka F, Lee L, Tamura I, Maekawa R, Aasada H, Yamagata Y, Sugino N. The role of melatonin as an antioxidant in the follicle. J Ovarian Res. 2012 Jan 26;5:5. doi: 10.1186/1757-2215-5-5. PMID 22277103
- [Background] Torres Fernandez ED, Huffman AM, Syed M, Romero DG, Yanes Cardozo LL. Effect of GLP-1 Receptor Agonists in the Cardiometabolic Complications in a Rat Model of Postmenopausal PCOS. Endocrinology. 2019 Dec 1;160(12):2787-2799. doi: 10.1210/en.2019-00450. PMID 31593246
- [Background] Voiculescu SE, Zygouropoulos N, Zahiu CD, Zagrean AM. Role of melatonin in embryo fetal development. J Med Life. 2014 Oct-Dec;7(4):488-92. PMID 25713608
- [Background] Williams T, Mortada R, Porter S. Diagnosis and Treatment of Polycystic Ovary Syndrome. Am Fam Physician. 2016 Jul 15;94(2):106-13. PMID 27419327
- [Background] Yesildaglar N, Yildirim G, Yildirim OK, Attar R, Ozkan F, Akkaya H, Yilmaz B. The effects of melatonin on endometriotic lesions induced by implanting human endometriotic cells in the first SCID-mouse endometriosis-model developed in Turkey. Clin Exp Obstet Gynecol. 2016;43(1):25-30. PMID 27048013
- [Background] Zegers-Hochschild F, Nygren KG, Adamson GD, de Mouzon J, Lancaster P, Mansour R, Sullivan E; International Committee Monitoring Assisted Reproductive Technologies. The ICMART glossary on ART terminology. Hum Reprod. 2006 Aug;21(8):1968-70. doi: 10.1093/humrep/del171. Epub 2006 Jul 24. PMID 16864610
- [Background] Zhang Y, Xu Y, Xue Q, Shang J, Yang X, Shan X, Kuai Y, Wang S, Zeng C. Discordance between antral follicle counts and anti-Mullerian hormone levels in women undergoing in vitro fertilization. Reprod Biol Endocrinol. 2019 Jul 4;17(1):51. doi: 10.1186/s12958-019-0497-4. PMID 31272468